CLINICAL TRIAL: NCT03276234
Title: Is There a Relationship Between Serum Sodium Level and Mean Platelet Volume (MPV) Value in Patients Undergoing Transurethral Prostate Resection (TUR)?
Brief Title: Is There a Relationship Between Serum Sodium Level and Mean Platelet Volume (MPV) Value
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-075
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Mean Platelet Volume According to Serum Sodium Value; on Patients Who Will Have Transurethral Resection of the Prostate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Is there a relationship between serum sodium level and mean platelet volume (MPV) value in patients undergoing transurethral prostate resection (TUR)?

DETAILED DESCRIPTION:
Thirty one patients undergoing transurethral prostate resection (TUR)? will be evaluated.The relationship between serum sodium value and MPV value of patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status 1 and 3
* Patients between the ages of 18 and 80

Exclusion Criteria:

* Patients with bleeding disorder
* Patients with blood transfusion
* Patients are that sodium values are lower than normal range.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients who will be done TUR.
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2017-09-13 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-11-29 (Estimated)

PRIMARY OUTCOMES:
Mean platelet volume | one month
  Changes in mean platelet volüme according to sodium value(Measurements of changes will be made twice in the study framework)

CONTACTS AND LOCATIONS:
Locations (1):
- Male patients between 18 and 80 years of age who have undergone TUR., Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided